CLINICAL TRIAL: NCT03578458
Title: Evaluation of a Novel Mobile Application to Assess Dietary Information
Brief Title: Novel Mobile Application to Assess Dietary Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17.13.NIHS
Record Dates: First submitted 2018-05-24; First posted 2018-07-06 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Dietary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- US Healthy diet (Other): Subjects will install a mobile app for use and will be randomly assigned to a healthy diet.
  Interventions: Other: subjects will install a mobile app for use
- Vegetarian diet (Other): Subjects will install a mobile app for use and will be randomly assigned to a vegetarian diet.
  Interventions: Other: subjects will install a mobile app for use
- Mediterranean diet (Other): Subjects will install a mobile app for use and will be randomly assigned to a Mediterranean diet.
  Interventions: Other: subjects will install a mobile app for use

INTERVENTIONS:
Other: subjects will install a mobile app for use — novel mobile application

SUMMARY:
The study will assess the accuracy of food capture methods using a novel mobile application. This will be done by comparing the energy and nutrient content of reported foods against those of foods actually consumed (i.e., reported vs actual). Two methods of using the application will be tested:

1. During each eating occasion to report foods and amounts consumed
2. By taking photographs of every food consumed, using the camera functionality of the mobile application and using the application the following day (according to the availability of the study subjects) to report foods and amounts consumed. This is to be consistent with the concept of a 24-hour dietary recall.

One group will use a standard 24-hour dietary recall method.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy men and women 18-65 years of age
* Eats a wide variety of foods from all food groups
* 18 ≤ body mass index (BMI) < 30 kg/m2
* Ability to read and write in English
* iPhone (iOS 11 or higher) or Android phone (6 or higher) user willing to download the mobile application

Exclusion Criteria:

* Presence of active disease at screening that would prevent normal dietary intake and/or would result in weight loss (irritable bowel syndrome, Crohn's disease, celiac disease, etc.)
* Medical complications or chronic illness that would prevent full participation (e.g., active cancer)
* Pregnant or lactating women
* Diagnosed eating disorder
* Vegetarian
* Special dietary requirements or severe allergies that prevent the consumption of major food groups (e.g., gluten free, lactose free, Halal)
* Diagnosis of a mental health condition that has not been stable within the past 6 months
* Current or previous experience with dietary data collection or analysis
* Concurrent participation in another research study at any point during the study
* Availability and access to a tablet device (iPad, Android) only
* Shift workers
* Plan to partake in vigorous physical training/ exercise during the study period (e.g., training for or running a marathon)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Energy and nutrient content captured on the mobile application | Day 1 intakes recorded on application after meals
  During each eating occasion to report foods and amounts consumed

SECONDARY OUTCOMES:
Energy and nutrient content captured on the mobile application by taking photographs of food consumed | Day 1 intakes photographed on application after meals
  During each eating occasion to report foods and amounts consumed
Assess whether food capture using the mobile application is comparable with a conventional 24-hour recall. | Day 1 intakes will be reviewed by recall method
  Use of application for food capture versus 24 hour dietary recall in reporting foods and amounts consumed

CONTACTS AND LOCATIONS:
Overall Officials: Sai Krupa Das, Ph.D, Principal Investigator — Tufts University USDA Human Nutrition Research Center on Aging (HNRCA), Boston MA
Locations (1):
- Tufts University USDA Human Nutrition Research Center on Aging (HNRCA), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blanchard CM, Chin MK, Gilhooly CH, Barger K, Matuszek G, Miki AJ, Cote RG, Eldridge AL, Green H, Mainardi F, Mehers D, Ronga F, Steullet V, Das SK. Evaluation of PIQNIQ, a Novel Mobile Application for Capturing Dietary Intake. J Nutr. 2021 May 11;151(5):1347-1356. doi: 10.1093/jn/nxab012. PMID 33693732